CLINICAL TRIAL: NCT04726150
Title: Effect of CoVid-19 and Exercise on Myocardial Fibrosis and Ventricular Arrhythmias (CovidEx)
Brief Title: Effect of CoVid-19 (CoronaVirusDisease-19) and Exercise on Myocardial Fibrosis and Ventricular Arrhythmias
Acronym: CoViDEx
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 1499
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2022-10

CONDITIONS: Covid19; Athletes Heart; Myocarditis Viral; Ventricular Arrythmia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood samples will be taken to determine the levels of hsTn
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mildly of Asymptomatic COVID: Athletes with prior COVID-19 that had a mildly or asymptomatic course
  Interventions: Other: ILR implantation
- Moderate to Severe Symptoms, Cardiac Symptoms: Athletes with prior COVID-19 that had a moderate to severely symptomatic course, or who experience(d) cardiac symptoms
  Interventions: Other: ILR implantation
- Hospitalized for: Athletes that were hospitalized for COVID-19
  Interventions: Other: ILR implantation

INTERVENTIONS:
Other: ILR implantation — If LGE is present on CMR, ILR implantation will be proposed

SUMMARY:
COVID-19 can cause myocarditis, which can cause myocardial fibrosis. This has been shown to increase mortality and morbidity among athletes. Several efforts have been made to guide sports participation after COVID-19, but not much scientific evidence is present to back-up those guidelines. The current initiative aims gain a heightened insight in this matter.To identify the presence of fibrosis athletes who recovered from COVID-19 will undergo CMR (Cardiac MRI). All athletes will also undergo echocardiography, 5-day Holtermonitoring among others. This will allow to determine whether differences between those with and those without fibrosis are present. If fibrosis is present, athletes will be offered an implantation of a very small monitoring device that will be able to detect arrhythmias with a much higher sensitivity. Also an exercise echocardiography will be performed, to determine the safety of continuation of athletic efforts.

Amendment:

Recently myocarditis and pericarditis have also been observed after the administration of mRNA-vaccines, specifically after the second dose. The effect of vaccination on exercise capacity is less clear. To investigate this we propose to amend the inclusion criteria for COVIDEX with "athletes undergoing or having undergone COVID vaccination"

DETAILED DESCRIPTION:
Baseline investigations will depend on the clinical presentation of the athlete. Three groups are identified:

1. Asymptomatic/mildly symptomatic: anosmia, ageusia, headache, mild fatigue, fever ≤3d, myalgias ≤3d , mild upper respiratory tract illness, and mild gastrointestinal illness
2. Moderate to severe symptoms: at least 2 of: persistent fever ≥4d, chills ≥4d, myalgias ≥4d, lethargy impairing activities of daily life (ADL) ≥4d, dyspnea during ADL ≥4d, and chest tightness ≥4d. Or cardiac symptoms: dyspnea, exercise intolerance, chest tightness, dizziness, (pre)syncope, and (new onset) palpitations.
3. Hospitalized: all athletes admitted for COVID-19, whether or not on the intensive care unit.

   * Group 1 will undergo a thorough history, clinical examination, ECG, laboratory tests for hs-Troponin T (TnT) and hsCRP, echocardiography at rest, 5-day-Holter and CMR. These examinations will take place at least 30 days after the first symptoms or positive test. Follow-up will be performed as pointed out with the grey crosses in the table. Depending on the results further investigation may be required (as in group 2 and 3). This part of the study is interventional in nature (not according to standard of care in those individuals).
   * Groups 2 and 3 will undergo a more extensive evaluation: a thorough history, clinical examination, ECG, laboratory tests for hs-TnT and hsCRP, echocardiography at rest, CardioPulmonary Exercise Test (CPET), 5-day-Holter, late potentials and CMR.

If in any athlete the CMR shows signs of fibrosis or myocarditis, an exercise echocardiography will be performed additionally. Those subjects will be part of a more extensive follow-up schedule (both white and grey in the table) In the case of the presence of a non-ischemic pattern of Late Gadolinium Enhancement (LGE) or raised myocardial T2 and normal of only mildly contractile reserve, implantation of an Implantable Loop Recorder (ILR) will be performed as a part of the study. This then will be remotely followed-up through telemonitoring. Other athletes (and those who refuse an ILR will receive a 5d-Holter monitoring.

Amendment:

Athletes having undergone complete vaccination will be asked to provide the investigators with their training data prior to and following boostervaccination. Those athletes undergo investigations already included in the COVIDEX study, albeit in a condensed manner (Ergospirometry, Echocardiography and Blood Sample). These tests will take place at the day before the second vaccination and seven days after. Those athletes will also be asked to provide the investigators with their training data prior to and following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Athletes (professional or recreational but aiming to compete at a national or international level), performing mixed-type or endurance sports as defined by Pelliccia et al. who:

  1. have recovered from a proven (either by PCR (Polymerase Chain Reaction), serology or chest Computed Tomography) COVID-19 infection
  2. are more than 1-month post onset of symptoms or the first positive PCR and
  3. are willing to start (or are) exercising again

Exclusion Criteria:

1. known prior cardiac fibrosis
2. known or newly diagnosed coronary artery disease
3. allergy or contraindications for gadolinium contrast.
4. unwillingness or impossibility to give informed consent
5. Presence of edema on the CMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Athletes >= 18 years if age who suffered from COVID, who are at least one month post diagnosis of COVID-19 and who are willing to start exercising again
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of athletes with LGE on CMR | 6months - 3 years post COVID diagnosis
Arrhythmic Burden on ILR | 6months to 2 to3 years post implantation (depending on device longevity)
Arrhythmic Burden on 5d Holter | At inclusion
Arrhythmic Burden on 5d Holter | At 6 months
Arrhythmic Burden on 5d Holter | At 12 months
Arrhythmic Burden on 5d Holter | At 3 years

SECONDARY OUTCOMES:
Occurrence of (pre)syncope or SCD | throughout the duration of the study, preamble is 3 years
Long-term evolution of cardiac function on echo/CMR: ejection fraction | reevaluation at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No